CLINICAL TRIAL: NCT01385046
Title: Project Fit:a School- and Community-based Intervention to Address Physical Activity and Healthy Eating Among Low-income Elementary School Children
Brief Title: Project Fit:a School- and Community-based Obesity Intervention
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Denise Holmes/Dean of Human Medicine, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSU-123
Record Dates: First submitted 2011-06-22; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
Keywords: physical inactivity; poor diet
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- physical activity and nutrition (Experimental)
  Interventions: Behavioral: Project Fit

INTERVENTIONS:
Behavioral: Project Fit — physical activity and nutrition education

SUMMARY:
Project FIT is a collaboration between the public school system, local health systems, physicians, neighborhood associations, businesses, faith-based leaders, community agencies and university researchers to develop a multi-faceted approach to promote physical activity and healthy eating toward the general goal of preventing and reducing childhood obesity among children in Grand Rapids, MI, USA. There are four overall components to Project FIT: school, community, social marketing, and school staff wellness - all that focus on: 1) increasing access to safe and affordable physical activity and nutrition education opportunities in the schools and surrounding neighborhoods; 2) improving the affordability and availability of nutritious food in the neighborhoods surrounding the schools; 3) improving the knowledge, self-efficacy, attitudes and behaviors regarding nutrition and physical activity among school staff, parents and students; 4) impacting the 'culture' of the schools and neighborhoods to incorporate healthful values; and 5) encouraging dialogue among all community partners to leverage existing programs and introduce new ones.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in participating school district in grades 1-5.

Exclusion Criteria:

* None

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by pedometer. | 2 years
  Physical activity will be measured with a pedometer worn for 7-day period at the beginning and end of the intervention.
Healthy eating index quantified by the Food Frequency Questionnaire. | 2 years
  The healthy eating index is a composite measure of diet quality.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Holmes, PhD, Study Chair — Michigan State University
Locations (1):
- Grand Rapids Public Schools, Grand Rapids, Michigan, United States

REFERENCES:
- [Derived] Eisenmann JC, Alaimo K, Pfeiffer K, Paek HJ, Carlson JJ, Hayes H, Thompson T, Kelleher D, Oh HJ, Orth J, Randall S, Mayfield K, Holmes D. Project FIT: rationale, design and baseline characteristics of a school- and community-based intervention to address physical activity and healthy eating among low-income elementary school children. BMC Public Health. 2011 Jul 29;11:607. doi: 10.1186/1471-2458-11-607. PMID 21801411
- See also: Related Info — http://www.theprojectfit.org/